CLINICAL TRIAL: NCT03005782
Title: A Phase 1, Open-Label, Dose-Escalation and Cohort Expansion First-in-Human Study of the Safety, Tolerability, Activity and Pharmacokinetics of REGN3767 (Anti-LAG-3 mAb) Administered Alone or in Combination With REGN2810 (Anti-PD-1 mAb) in Patients With Advanced Malignancies
Brief Title: Study of REGN3767 (Anti-LAG-3) With or Without REGN2810 (Anti-PD1) in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3767-ONC-1613; 2016-002789-30 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-12-29 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Malignancies
MeSH Terms: conditions — Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy (REGN3767) (Experimental): Group A will consist of up to 4 sequential dose cohorts. Each cohort will receive 1 of 3 ascending dose levels of study drug during dose escalation. In addition 1 tumor-specific cohort will be treated at the recommended phase 2 dose (RP2D) during dose expansion.
  Interventions: Drug: REGN3767
- Combination Therapy (REGN3767+cemiplimab) (Experimental): Group B will consist of up to 4 sequential dose cohorts. Each cohort will receive 1 of 3 ascending dose levels of study drug during dose escalation. In addition, 9 tumor-specific cohorts will be treated at the RP2D during dose expansion
  Interventions: Drug: REGN3767; Drug: cemiplimab

INTERVENTIONS:
Drug: REGN3767
  Other Names: fianlimab
Drug: cemiplimab
  Other Names: REGN2810
  Arms: Combination Therapy (REGN3767+cemiplimab)

SUMMARY:
The primary objectives in the dose escalation phase are to evaluate safety and pharmacokinetics (PK) in order to determine the selected dose level(s) for expansion of REGN3767 as monotherapy and in combination with cemiplimab in patients with advanced malignancies, including lymphoma.

The primary objectives in the dose expansion phase are to assess preliminary anti-tumor activity of REGN3767 alone and in combination with cemiplimab (separately by cohort) as measured by objective response rate (ORR).

ELIGIBILITY:
Key Inclusion Criteria:

* Dose escalation cohorts: Patients with histologically or cytologically confirmed diagnosis of malignancy (including lymphoma) with demonstrated progression of a tumor for whom there is no available therapy likely to convey clinical benefit AND who have not been previously treated with a PD-1/PD-L1 inhibitor. These patients do not require measurable disease
* Dose expansion cohorts: Patients with histologically or cytologically confirmed diagnosis of 1 of specified tumors with measurable disease per RECIST 1.1 or Lugano criteria. Some patients may have been previously treated with a PD-1 or PD-L1 inhibitor
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate organ and bone marrow function

Key Exclusion Criteria:

* Prior treatment with any LAG-3 targeting biologic or small molecule
* Radiation therapy within 2 weeks prior to randomization and not recovered to baseline from any AE due to radiation
* Untreated or active central nervous system metastases - Ongoing or recent (within 5 years) evidence of significant autoimmune disease
* Corticosteroid therapy (>10 mg prednisone/day or equivalent) within 1 week prior to the first dose of study drug
* Myocardial infarction within 6 months

Note: Other protocol defined Inclusion / Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (Dose Escalation Phase) | Baseline to 28 days
Rate of adverse events (Dose Escalation Phase) | Baseline to 51 weeks
Rate of serious adverse events (Dose Escalation Phase) | Baseline to 51 weeks
Occurrence of death (Dose Escalation Phase) | Baseline to 51 weeks
Number of patients with laboratory abnormalities (grade 3 or higher per Common Terminology Criteria for Adverse Events [CTCAE]) (Dose Escalation Phase) | Baseline to 51 weeks
Area under the curve (AUC) computed from time zero to the time of the last concentration [AUCall] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
AUCall-to-dose ratio [AUCall/Dose] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
AUC from time zero extrapolated to infinity [AUCinf] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
AUCinf-to-dose ratio [AUCinf/dose] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
AUC computed from time zero to the time of the last positive concentration [AUClast] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
AUClast-to-dose ratio [AUClast/dose] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Clearance [CL] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Maximum Plasma Concentration [Cmax] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to week 51
Cmax-to-dose ratio [Cmax/dose] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Last positive (quantifiable) concentration [Clast] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Mean residence time extrapolated to infinity [MRTinf] (Dose Escalation Phase) | Baseline to 51 weeks
Mean residence time when the drug concentration profile is based on values up to and including the last positive concentration [MRTlast] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Observed terminal half-life [t1/2] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
t1/2 beta (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Time of the last positive (quantifiable) concentration [tlast] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Time to Cmax [tmax] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Volume of distribution at steady state [Vss] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Volume of distribution of the terminal phase [Vz] (Primary: Dose Escalation Phase; Secondary: Dose Expansion Phase) | Baseline to 51 weeks
Objective response rate based on RECIST 1.1 for Solid Tumors (Dose Expansion phase) | Baseline to 51 weeks
Objective response rate by Lugano criteria for Lymphoma (Dose Expansion Phase) | Baseline to 51 weeks

SECONDARY OUTCOMES:
Objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (solid tumors) (Dose Escalation Phase) | Baseline to week 51
Objective response rate per Lugano criteria (lymphomas) (Dose Escalation Phase) | Baseline to week 51
Best overall response based on RECIST 1.1 criteria (Dose Escalation Phase) | Baseline to 51 weeks
Best overall response based on irRECIST criteria (Dose Escalation Phase) | Baseline to 51 weeks
Best overall response based on Lugano criteria (Dose Escalation Phase) | Baseline to 51 weeks
Duration of response based on RECIST criteria (Dose Escalation Phase) | Baseline to week 51
Duration of response based on irRECIST criteria (Dose Escalation Phase) | Baseline to week 51
Duration of response based on Lugano criteria (Dose Escalation Phase) | Baseline to week 51
Disease control rate based on RECIST criteria (Dose Escalation Phase) | Baseline to 51 weeks
Disease control rate based on irRECIST criteria (Dose Escalation Phase) | Baseline to 51 weeks
Disease control rate based on Lugano criteria (Dose Escalation Phase) | Baseline to 51 weeks
Progression free survival based on RECIST (Dose Escalation Phase) | Baseline to 51 weeks
Progression free survival based on irRECIST (Dose Escalation Phase) | Baseline to 51 weeks
Progression free survival based on Lugano criteria (Dose Escalation Phase) | Baseline to 51 weeks
Incidence of adverse events (Dose Expansion Phase) | Baseline to 51 weeks
Incidence of serious adverse events (Dose Expansion Phase) | Baseline to 51 weeks
Incidence of death (Dose Expansion Phase) | From Baseline to the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 42 months
Number of patients with laboratory abnormalities (grade 3 or higher per Common Terminology Criteria for Adverse Events [CTCAE]) (Dose Expansion Phase) | Baseline to 51 weeks
Incidence of anti-drug antibodies (Dose Escalation Phase and Dose Expansion Phase) | Baseline to 51 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (43):
- United States (33):
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - California Cancer Associates For Research And Excellence, Fresno, California
  - University of California San Diego (UCSD), La Jolla, California
  - The Angeles Clinic, Los Angeles, California
  - University of California Davis Health Systems, Sacramento, California
  - California Pacific Medical Center (CPMC), San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Lombardi Comprehensive Cancer Center - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Dana Farber Cancer Institute, Jamaica Plain, Massachusetts
  - Henry Ford Health Hospital, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Washington University in Saint Louis, St Louis, Missouri
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Cancer Care Alliance-UNM Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health-Monter Cancer Center, Lake Success, New York
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University Hospitals Seidman Cancer Center and Case Western Reserve University, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Virginia Cancer Care Specialist, PC, Fairfax, Virginia
- Australia (3):
  - The University of Western Australia - The Queen Elizabeth II Medical Centre (QEIIMC) - Sir Charles Gairdner Hospital (SCGH), Perth, Western Australia
  - Royal Brisbane and Women's Hospital, Brisbane
  - Peter Maccallum Cancer Centre (PMCC), Melbourne
- St. Vincents University Hospital, Dublin, Ireland
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- United Kingdom (2):
  - Guy's Hospital, London, Europe
  - University Of Oxford - Churchill Hospital, Headington, Oxford

REFERENCES:
- [Derived] Hamid O, Lewis KD, Weise A, McKean M, Papadopoulos KP, Crown J, Kim TM, Lee DH, Thomas SS, Mehnert J, Kaczmar J, Lakhani NJ, Kim KB, Middleton MR, Rabinowits G, Spira AI, Yushak M, Mehmi I, Fang F, Chen S, Mani J, Jankovic V, Wang F, Fiaschi N, Brennan L, Paccaly A, Masinde S, Salvati M, Fury MG, Kroog G, Lowy I, Gullo G. Phase I Study of Fianlimab, a Human Lymphocyte Activation Gene-3 (LAG-3) Monoclonal Antibody, in Combination With Cemiplimab in Advanced Melanoma. J Clin Oncol. 2024 Aug 20;42(24):2928-2938. doi: 10.1200/JCO.23.02172. Epub 2024 Jun 20. PMID 38900987